CLINICAL TRIAL: NCT03019471
Title: Non Invasive Cancer Test (NICT): a Proof of Principle Study.
Acronym: NICT-NIPT-CA
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL55080.068.15
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-05

CONDITIONS: Neoplasmata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Lung cancer: Isolate Tumor DNA from the patients blood.
  Interventions: Genetic: Isolation of tumor DNA
- Breast cancer: Isolate Tumor DNA from the patients blood.
  Interventions: Genetic: Isolation of tumor DNA
- Colorectal cancer: Isolate Tumor DNA from the patients blood.
  Interventions: Genetic: Isolation of tumor DNA
- Glioma: Isolate Tumor DNA from the patients blood.
  Interventions: Genetic: Isolation of tumor DNA

INTERVENTIONS:
Genetic: Isolation of tumor DNA

SUMMARY:
The investigators aim to collect tumor DNA out of blood of cancer patients. If this is successful this could lead to the development of a cancer test in blood in the future, which is less invasive than current diagnostic methods.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed local or metastatic breast cancer, colorectal cancer, non-small cell lung cancer and anaplastic glioblastoma, before start of radiation therapy, chemoradiation or chemotherapy.
2. Patients age > 18 years, willing and able to comply with the protocol as judged by the investigator with a signed informed consent

Exclusion Criteria:

1. Patients with a history of malignant disease other than the disease under study, with an exception for adequately treated squamous cell carcinoma of the skin, basal cell carcinoma of the skin and in situ cervix carcinoma.
2. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with newly diagnosed local or metastatic breast cancer, colorectal cancer, non-small cell lung cancer and anaplastic glioblastoma, before start of radiation therapy, chemoradiation or chemotherapy.
  2. Patients age > 18 years, willing and able to comply with the protocol as judged by the investigator with a signed informed consent
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ctDNA | One year
  Demonstrate the presence or absence of ctDNA in patients plasma. Examine if there us a sufficient concentration of ctDNA in the plasma to reliably diagnose cancer and determine the CNV

CONTACTS AND LOCATIONS:
Overall Officials: Christine C. De Die-Smulders, Prof. dr., Principal Investigator — Clinical Geneticist in MUMC+
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No